CLINICAL TRIAL: NCT00711438
Title: Phase II Pilot Pragmatic Single-Blinded Fast Track Randomised Controlled Trial of the Breathlessness Intervention Service Versus Standard Care for Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Pilot Randomized Controlled Trial of a Breathlessness Intervention Service for Chronic Obstructive Pulmonary Disease
Acronym: BIS-PhIInm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Dr Sara Booth, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BIS PhIInm v3 26/10/06
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2006-10

CONDITIONS: Dyspnea
Keywords: Breathlessness; Dyspnoea; Dyspnea; Palliative care; RCT; Randomised controlled trial; COPD; Chronic respiratory disease
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FT (Experimental): Breathlessness Intervention Service (BIS)
  Interventions: Behavioral: Breathlessness Intervention Service (BIS)
- WL (Active Comparator): Best supportive care
  Interventions: Behavioral: Best supportive care (Standard care)

INTERVENTIONS:
Behavioral: Breathlessness Intervention Service (BIS) — BIS consists of a clinical specialist physiotherapist & palliative care consultant. It aims to manage the symptom of breathlessness in patients with any disease using a rehabilitative approach. Interventions include: evidence-based non-pharmacological interventions (psychological, social & physical); palliative care input (e.g. end of life issues, psychosocial issues, family concerns); & pharmacological review. This BIS seeks to enhance self-management of breathlessness. Uniquely, care is located in clinic or in patients' own homes, as appropriate. Referrals come from medical specialists, GPs & allied health professionals (with medical consent).
  Other Names: BIS
  Arms: FT
Behavioral: Best supportive care (Standard care) — Standard care: specialist outpatient appointments in secondary care (e.g. respiratory) which may include specialist nurse input, and primary care services.
  Other Names: Standard care
  Arms: WL

SUMMARY:
The aim of this study is to test the feasibility of conducting a pragmatic fast track Randomized Controlled Trial (RCT) of the Breathlessness Intervention Service (BIS) versus standard care for patients with COPD and their carers, and to begin testing the effectiveness of the intervention.

DETAILED DESCRIPTION:
The aim of the study is to test the feasibility of conducting a pragmatic single-blinded fast track RCT of BIS versus standard care for patients with COPD and their carers and to begin testing the effectiveness of the intervention by: (1) Describing the referral patterns and activity of the service; (2) Describing the experiences and views of the service by people with breathlessness who have been referred to it and the experiences and views of those informally involved in their care; (3) Identifying those aspects of the service which are most useful to people with breathlessness, those informally involved in their care and health care professionals.

The study consists of five components: (1) data relating to referral patterns and service activity; (2) identification of components of the intervention; (3) a pilot pragmatic fast-track randomised controlled trial (RCT) of BIS for COPD patients versus standard care; (4) semi-structured interviews with referrers; (5) in-depth interviews with BIS staff. The RCT is described below.

Although the BIS also receives referrals for patients with cancer and heart failure, COPD patients make up the largest diagnostic group of referrals. The pilot trial therefore focuses on a heterogeneous cohort of COPD/COAD patients.

The investigator will be blinded to the allocation of respondents until week 8. This will be achieved by the investigator conducting the recruitment to the study and collecting baseline measures, but then passing the process of randomisation and reporting of allocation (to the patient and provider) over to a third party (clinical trials' nurses) using a random sequence of opaque envelopes previously generated by a study administrator at King's (independent of the service and the RCT). Subsequent to this, all data will be handled using study identity numbers and group allocation identifiers will only be added at the analysis stage. Outcomes are all self-assessed by patients and carers principally using structured questionnaires but also incorporating a qualitative topic guide prior to randomisation and then again at the end of the fast track group's exposure to BIS and the control group's waiting period for BIS (at both of these measurement points structured questionnaires will be completed prior to the qualitative interview).

Subsequent data collected from the control group once they are in receipt of BIS (after their period on the waiting list when their group allocation was blinded to the investigator) will be treated as before/after data and not RCT data. This will allow the collection of qualitative data at the midpoint of using the service as the investigator will no longer be blinded to their group allocation, nor will she be required to be at this stage.

Measurement points: 'measures' (quantitative and qualitative) will be taken for all respondents (FT and CC) at baseline (t1), prior to randomisation. They will be repeated for the fast-track group (FC) during the intervention (4 weeks post commencement of the intervention (FTt2) - quantitative only) and for control condition group at the same time (CCt2 - quantitative only), and then again after discharge for the fast track group (8 weeks post commencement of intervention (FTt3)). As well as being measured at t1 (randomisation) and t2 (mid-point between randomisation and intervention - quantitative only), the control condition group (CC) will also be measured just prior to the commencement of their intervention (CCt3), repeated during the intervention (4 weeks post commencement of the intervention (CCt4)) and then again after discharge (8 weeks post commencement of intervention (CCt5)). Using this measurement strategy should make it possible to identify whether or not the condition of respondents in the control group deteriorated whilst they awaited their intervention and whether or not this then had an impact on final outcomes for this group.

Measures will be collected by means of audio-taped structured/semi-structured interviews (with respondents' permission). It is proposed that at each measurement point patients and carers are interviewed separately as this found to be important in the pilot study interviews. This will be managed by means of requesting that carers complete any self-complete measures whilst the interview is being conducted with the patient. Interviews with carers will then be conducted on a separate, but temporally close, occasion (e.g. up to 2 days later), at the carer's convenience (e.g. in the evening if required). Careful attention will be paid to the needs of the patient and carer in terms of fatigue.

Determining the sample size for a pilot/exploratory trial of this type is difficult. As no trials have been conducted before with this particular intervention, or for this type of intervention with this patient group (i.e. COPD patients), there is a lack of data (e.g. identification of primary outcome measures and their data) to support the power calculations usually used to estimate the required sample size of a definitive RCT (i.e. the number of participants needed to ensure the study is scientifically sound). In addition, those trials that do exist relating to interventions for patients with COPD (e.g. trials of pulmonary rehabilitation rather than breathlessness intervention services) have focused primarily on physiological outcomes such as clinical measures of breathlessness. However, as a result of our earlier work at the Pre-Clinical phase and Phase I, we became aware of the need to look beyond such physiological measures and consider other outcomes (e.g. distress due to breathlessness, ability to choose to participate in social events).

Thus the pilot/exploratory trial (Phase II) will itself provide vital information to inform the power calculations for a future planned definitive RCT (Phase III). The aims of this current pilot/exploratory trial therefore include testing the intervention (the BIS) but also establishing the feasibility of conducting a definitive RCT by testing the trial method (i.e. the pragmatic fast-track design), randomisation procedures and the identification of appropriate primary outcome measures. It is envisaged that the most likely primary patient outcomes will be 'distress due to breathlessness' and mastery of breathlessness; the most likely primary carer outcome is 'carer distress due to breathlessness'. For both patients and carers 'distress due to breathlessness' will be measured using a Visual Analogue Scale (VAS; 0-10cm); a difference between the baseline and follow up measurements of 1cm on this scale could be regarded as clinically significant for patients with intractable breathlessness. This pilot/exploratory RCT will provide the data to confirm or refute these outcomes, and so enhance the design of future definitive trials.

Based on clinical experience, data published from other studies and case reports (e.g. Corner et al, 1996), and on expert advice, we have made some tentative estimates of the likely changes we may expect the intervention to have. We could expect a change in score of severe distress due to breathlessness of 2.2 (SD 1.8) on a 10 point scale. This difference would be detected, using a Mann Whitney U test, with 11 patients in each group (22 in total), with 80% power and a significance of p=0.05. A change in the proportion of patients with severe or very severe distress due to breathlessness from 90% to 40% would be detected at 80% power and a significance of p<0.05 by 14 patients in each group (28 patients in total). Therefore we will aim to recruit at least 30 (or 28) patients to the trial.

A number of subjective measures, exercise tolerance measures and physiological measures are already collected or recorded by the BIS itself (e.g. VAS, modified BORG, MRC grading of dyspnoea symptoms etc.). These will continue to be collected and will be utilised by both the service and the evaluation. In accordance with the aims of the evaluation, other outcomes to be assessed within the trial will relate to patient and carer satisfaction with the service, patient and carer quality of life, patient and carer anxiety, patient mastery, caregiver burden, patients' breathlessness, patient and carer distress due to breathlessness, aspects of the service most useful to users (patients and carers) and other service use.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Appropriate referral to the BIS
* Diagnosis of COPD/COAD
* Aged 18 years or over
* Any patient who does not meet any of the exclusion criteria

Carers:

* The informal carers of patients specified above, who can be significant others, relatives, friends or neighbours
* Aged 18 years or over
* Any carer who does not meet the exclusion criteria

Exclusion Criteria:

* Any patient/carer unable to give informed consent
* Any patient living outside of Cambridgeshire PCT, West Essex PCT, East & North Hertfordshire PCT, or Suffolk PCT
* Any patient who has previously had access to BIS
* Any patient/carer who is demented or confused
* Any patient/carer with learning difficulties
* Any patient/carer from other vulnerable groups (e.g. head injury, severe trauma, and mental illness)
* Any patient/carer who does not meet all of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) - distress due to breathlessness | End of intervention (8 weeks after baseline)

SECONDARY OUTCOMES:
Modified BORG | As for primary outcome measure
VAS breathlessness at best /worst | As for primary outcome measure
Mastery scale of CRQ | As for primary outcome measure
SEIQoL-DW | As for primary outcome measure
HADS | As for primary outcome measure
social functioning | As for primary outcome measure
WHO Performance scale | As for primary outcome measure
experience of breathlessness & expectations / views of BIS | As for primary outcome measure
Carer Burden Interview and Caregiver Appraisal Scale | As for primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Sara Booth, FRCP, Principal Investigator — Cambridge University Hopsitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Booth S, Silvester S, Todd C. Breathlessness in cancer and chronic obstructive pulmonary disease: using a qualitative approach to describe the experience of patients and carers. Palliat Support Care. 2003 Dec;1(4):337-44. doi: 10.1017/s1478951503030499. PMID 16594223
- [Background] Booth S, Farquhar M, Gysels M, Bausewein C, Higginson IJ. The impact of a breathlessness intervention service (BIS) on the lives of patients with intractable dyspnea: a qualitative phase 1 study. Palliat Support Care. 2006 Sep;4(3):287-93. doi: 10.1017/s1478951506060366. PMID 17066970
- [Background] Booth S, Wade R. Oxygen or air for palliation of breathlessness in advanced cancer. J R Soc Med. 2003 May;96(5):215-8. doi: 10.1177/014107680309600503. No abstract available. PMID 12724429
- [Background] Booth S, Adams L. The shuttle walking test: a reproducible method for evaluating the impact of shortness of breath on functional capacity in patients with advanced cancer. Thorax. 2001 Feb;56(2):146-50. doi: 10.1136/thorax.56.2.146. PMID 11209105
- [Background] Booth S. The management of dyspnoea in advanced cancer. Hosp Med. 1998 May;59(5):348-9. No abstract available. PMID 9722382
- [Background] Bausewein C, Farquhar M, Booth S, Gysels M, Higginson IJ. Measurement of breathlessness in advanced disease: a systematic review. Respir Med. 2007 Mar;101(3):399-410. doi: 10.1016/j.rmed.2006.07.003. Epub 2006 Aug 17. PMID 16914301
- [Background] Bausewein C, Booth S, Gysels M, Higginson I. Non-pharmacological interventions for breathlessness in advanced stages of malignant and non-malignant diseases. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD005623. doi: 10.1002/14651858.CD005623.pub2. PMID 18425927
- [Background] Booth S, Wade R, Johnson M, Kite S, Swannick M, Anderson H; Expert Working Group of the Scientific Committee of the Association of Palliative Medicine. The use of oxygen in the palliation of breathlessness. A report of the expert working group of the Scientific Committee of the Association of Palliative Medicine. Respir Med. 2004 Jan;98(1):66-77. doi: 10.1016/j.rmed.2003.08.008. PMID 14959816
- [Derived] Farquhar MC, Higginson IJ, Fagan P, Booth S. The feasibility of a single-blinded fast-track pragmatic randomised controlled trial of a complex intervention for breathlessness in advanced disease. BMC Palliat Care. 2009 Jul 7;8:9. doi: 10.1186/1472-684X-8-9. PMID 19583857